CLINICAL TRIAL: NCT04988529
Title: A Pilot Randomized Control Trial Investigating the Effect of a Smartphone-based Serious Game on Depressive Symptoms.
Brief Title: Investigating the Effect of a Smartphone-based Serious Game on Depressive Symptoms.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Jaume I (Other)
Collaborators: Conselleria de Innovación, Universidades, Ciencia y Sociedad Digital. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SERGAMIN/278
Record Dates: First submitted 2021-07-09; First posted 2021-08-03 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone-based supported serious game intervention (Experimental): Group that receives the smartphone-based serious game intervention and receives technical support
  Interventions: Behavioral: Smartphone-based serious game intervention
- Waiting list control (No Intervention): Group that does not receive any treatment

INTERVENTIONS:
Behavioral: Smartphone-based serious game intervention — Smartphone-based serious game intervention consists in the use of a serious game designed specifically to improve depressive symptoms. The psychological content consists of CBT intervention with the following psychotherapeutic components: Motivation for change, Psychoeducation, Cognitive Flexibility, Behavioural Activation, and positive psychotherapeutic strategies. To encourage physical activity, the serious game incorporates a mixed reality through physical activities such as taking a walk in real life affects aspects inside the game.
  Arms: Smartphone-based supported serious game intervention

SUMMARY:
The objective of the present project is to study the effect of a smartphone-based serious game intervention for depressive symptoms. The serious game is based on Cognitive Behavior Therapy CBT, being behavioural activation and the promotion of physical activity one of the most important components.

DETAILED DESCRIPTION:
Due to the current COVID-19 pandemic and the effects of quarantine on people's daily lives, a dramatic increase in people suffering from symptoms of depression is expected; one of the most common mental disorders globally, the primary cause of suicide deaths in Europe and the major contributor to the overall global burden of disease.

Although there are effective treatments for depression, more than half of those affected worldwide (and more than 90% in many countries) do not receive these treatments. The dominant model of treatment delivery (individual face-to-face therapy) will not be enough to reach the majority of people who need treatment. Hence, one of the most important challenges within this scope is the design of new forms of treatment delivery to maximize the efficacy and dissemination of psychological treatment.

The use of the Information and Communication Technologies (ICTs) has allowed a new effective ways of treatment, endorsed by several studies; and the use of serious video games as a partial or complete form of treatment, whose own characteristics make them potentially effective for the treatment of mental health, has opened the possibility of a still very new field of study. The arrival of smartphones has increased the possibilities of designing online therapies for mental health and facilitated the use of games as therapy.

Therefore, the objective of the present project is to study the effect of a smartphone-based serious game intervention for depressive symptoms through a two armed pilot randomized control trial. A minimum of 40 participants diagnosed with mild to moderate depression symptoms will be randomly assigned to one of the two experimental conditions: a smartphone-based serious game condition, and a waiting list control condition. The researchers' hypothesis is that the smartphone-based serious game intervention will produce a significant improvement in depressive, anxious symptomatology and improved well-being after treatment compared to the waiting list control group.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Being able to read and understand Spanish
* Being able to use a smartphone
* Having an Android smartphone with internet connection
* Suffering from mild to moderate depressive symptoms (from 14 to 28 on the Beck Depression Inventory-II [BDI-II]

Exclusion Criteria:

* Suffering a severe mental disorder: bipolar disorder, alcohol and/ or substance dependence disorder, psychotic disorder, or dementia
* Having a high suicide risk (ideation or plan assessed by the MINI and item 9 of the BDI-II)
* Receiving another psychological treatment while the study is still ongoing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Up to 12 months
  The PHQ-9 is the depression module of the self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 consists of 9 items ranging from "0" (not at all) to "3" (nearly every day). It has a dual-purpose instrument since it can establish both depressive disorder diagnoses and grade depressive symptom severity. Scores can range from zero to 27. Scores of 15 or greater indicated major depression.
Beck Depression Inventory (BDI-II) | Up to 12 months
  The BDI-II is widely used to detect and assess the severity of depressive symptoms. The BDI-II consists of 21 multiple-choice items ranging from 0 to 3. It covers the different symptoms of major depression disorder in the DSM-IV. Scores can range from zero to 63. Scores greater than 29 mean major depression. The BDI-II has high internal consistency (alpha = 0.76 to 0.95) and for the Spanish version (alpha = 0.89) (Sanz, 2003)
Positive and negative emotionality Positive and Negative Affect Scale (PANAS) | Up to 12 months
  The PANAS is used to measure trait and state affectivity. The PANAS consists of 20 items divided in two independent 10-item dimensions to assess positive affect (PA) and negative affect (NA). Each item rated on a 5-point Likert-type scale. Low levels of PA predict the onset depreesion, reduce positive emotions, and increase the severity of depressive symptoms.Patients with more comorbid diagnoses had significantly higher NA and lower PA. It is brief, reliable, and has shown excellent internal consistency (alpha = 0.84 to 0.90) and convergent and divergent validity. The Spanish version has also shown high internal consistency (alpha = 0.87 and 0.89 for PA and NA in men, respectively, and alpha = 0.89 and 0.91 for PA and NA in women, respectively (Díaz-García, 2020).
Overall Anxiety Severity and Impairment Scale (OASIS) | Up to 12 months
  The OASIS is used to assess the severity and frequency of anxiety symptoms. Moreover, the scale provides information about behavioral avoidance and functional impairments in pleasurable activities, work, school or social relationship interference related to these symptoms in the last week. The OASIS consists of a 5-item self-report measure rated from 0 to 4 and are summed to obtain one total score. OASIS score of 8 or above would be indicative of a probable anxiety disorder. It has demonstrated strong psychometric properties with good internal consistency (alpha = 0.86), as well as test-retest reliability (K = 0.82) and convergent validity (Norman, 2006; Campbell-Sill, 2009; Norman, 2011).
Overall Depression Severity and Impairment Scale (ODSIS) | Up to 12 months
  The ODSIS is used to assess the severity and frequency of depressive symptomatology and functional deficits in pleasurable activities due to the depressive symptomatology. The ODSIS consists of a 5-item self-report measure rated from 0 to 4 with higher scores indicating greater depression-related severity and impairment. It has excellent internal consistency (alpha = 0.92) and it shows good convergent/discriminant validity (Bentley, 2014) Spanish version will be used (Mira, 2019

SECONDARY OUTCOMES:
System Usability Scale (SUS) | Up to 12 months
  he SUS is used to measure the usability of a software collecting the user's opinion. The SUS consists of a questionnaire of 10 items with 5 answer options rated from "o" (strongly disagree) to "4" (strongly agree)is a brief, reliable scale for measuring the usability of a program. It consists of a 10-item questionnaire with 5 response options, from 0 ("strongly disagree") to 4 ("strongly agree"). It could indicate that the user has had technical difficulties with the program. The Spanish version has been used in several research studies (Botella, 2016; Campos, 2018) and its validation process is currently ongoing.
Expectation of treatment scale and opinion of treatment scale (CEQ) | Up to 12 months
  (Devilly & Borkovec, 2000). The CEQ is a quick and easy-to-administer scale used to measure treatment expectations before the intervention and the satisfactions after the receiving intervention. Both instruments consist of 6 items rated from "0" (not at all) to 10 ("very much"). The Spanish version has been used in previous studies (Botella 2016; Mira, 2019; Tortella-Feliu, 2011)

CONTACTS AND LOCATIONS:
Locations (1):
- University Jaume I, Castellon, Castelló, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about GEOTEC, the technical research group of the University Jaume I — http://geotec.uji.es/
- See also: Information about the Laboratory of Psychology and Technology of the University Jaume I — http://www.labpsitec.uji.es/esp/index.php